CLINICAL TRIAL: NCT03567343
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Effects of a Proprietary Spearmint Extract Blend, on Sleep in Healthy Men and Women
Brief Title: Investigational Test of a New Sleep Supplement
Acronym: InTeNSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Kemin Foods LC (Industry)
Responsible Party: Principal Investigator, MICHAEL A GRANDNER, Assistant Professor of Psychiatry, Psychology, and Medicine Director, Sleep & Health Research Program, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1803377507
Record Dates: First submitted 2018-05-16; First posted 2018-06-25 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-02

CONDITIONS: Sleep; Mood; Cognitive Performance
Keywords: sleep

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprietary Spearmint Extract Blend (Active Comparator): Subjects randomized into the active treatment group will be asked to consume 500 mg/day of the Proprietary Spearmint Extract Blend blend by mouth every night 30 mins before bed, complete a sleep diary upon waking and wear a Fitbit Charge 2 device for sleep monitoring for 30 days.
  A subset of this group will undergo 2 overnight polysomnography studies
  Interventions: Dietary Supplement: Proprietary Spearmint Extract Blend
- Control (Placebo Comparator): Subjects randomized into the active treatment group will be asked to consume 500 mg/day of the excipient, microcrystalline cellulose by mouth every night 30 mins before bed, complete a sleep diary upon waking and wear a Fitbit Charge 2 device for sleep monitoring for 30 days.
  A subset of this group will undergo 2 overnight polysomnography studies
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Proprietary Spearmint Extract Blend — Water extracted spearmint extract and green tea blend
  Arms: Proprietary Spearmint Extract Blend
Other: Control — Placebo
  Arms: Control

SUMMARY:
This study seeks to observe the effects of a proprietary spearmint extract and green tea blend on sleep quality and duration. The study observes the effect of the supplement regarding sleep quality, and mental health.

DETAILED DESCRIPTION:
Sleep disturbance is common in adults and when it persists may result in chronic disease, excess health care utilization, mental disorders, health-risk behaviors, limitations of daily functioning, lost productivity, injury, and mortality (IOM 2006). An estimated 50-70 million adults in the United States have chronic sleep and wakefulness disorders (IOM 2006; Ram 2010) and many more adults report insufficient or deprived sleep. Data from 2014 indicates that approximately 35% of the US population is receiving insufficient sleep (Liu et al., 2016). This is alarming, since insufficient sleep is associated with cardiometabolic disease risk factors including weight gain, obesity, hypertension, diabetes, and inflammation (Grandner et al., 2016), as well as poor daytime functioning and many other outcomes (Grandner, 2017). Cognitive deficits are routinely seen in the laboratory, especially on the Psychomotor Vigilance Task (PVT) (Lim and Dinges, 2010). The National Institutes of Health suggests that adults aim for 7-8 h of sleep per night; however, approximately 28% of adults in the United States reported sleeping 6 h or less based on data from 2008 to 2010 (Schoenborn 2010).

A number of strategies are recommended to promote sleep quality and quantity, including a series of behavioral recommendations, such as keeping to a routine sleeping schedule, the timing of eating and physical activity in relation to bedtime, avoidance of stimulants, and maintaining a bedroom environment conducive to sleep (National Sleep Foundation 2015). Although, pharmacologic options are available to treat sleep disturbances, there is consumer interest in natural sleep remedies due to concerns with side effects, dependency, and the safety of prescription medications. The current study seeks observe the effects of a new proprietary blend containing spearmint and green tea extract. It will be the first randomized, double-blind, placebo controlled trial observing the effects of 30 days of 500 mg of a blend containing Spearmint extract and green tea on sleep when administered 30 minutes before bed. This study will utilize Fit-bit (San Francisco, California) (a tool whose use for evaluation of sleep is growing) for daily evaluation of sleep throughout the study in addition to polysomnography, considered by many researchers to be the gold standard for evaluation of sleep outcomes, at chosen timepoints.

ELIGIBILITY:
INCLUSION CRITERIA

To be included in the study, patients must:

1. Subject is a male or female, 22-50 years of age, inclusive.
2. Subject is judged by the Investigator to be in general good health on the basis of medical history.
3. Subject is a non-user of nicotine products for 6 months prior to screening.
4. Subject's initial online screen reveals a score >5 on the PSQI.
5. Subject has a BMI of 18.50-29.99 kg/m2, inclusive, at screening.
6. Subject is willing to maintain habitual diet and activity patterns throughout the study period, other than the study instructions given for caffeine, alcohol, and vigorous physical activity.
7. Subject is willing to consume study product 30 minutes before bed throughout the study period.
8. Subject will consume no more than 14 alcoholic drinks (12oz beer, 5oz wine, 1.5oz distilled spirits) per week while in the study, no more than 4 drinks on a single occasion, and no more than 1 alcoholic drink within 4 hours of bedtime.
9. Subject will consume no more than 4 servings of caffeine substances per day (8oz coffee, 1oz espresso, 12oz caffeinated soda, 8oz energy drink) and no caffeine within 6 hours of bedtime.
10. Subject will refrain from vigorous physical activity (causing sweating) within 2 hours of bedtime.
11. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

EXCLUSION CRITERIA

1. Subject has a history or presence of clinically important cardiac, renal, hepatic, endocrine, pulmonary, biliary, pancreatic, chronic pain condition(s), or neurologic disorders.
2. Subject has a history of diagnosed clinical depression in the prior 2 years of screening. This will be determined by self report at screening (PHQ9 scores indicating likely depression diagnosis (<=2 on items 1 or 2, plus <=2 on at least 5 other symptoms) will be exclusionary) and with the Mini International Neuropsychiatric Inventory assessed at the screening visit.
3. Subject has an active infection or signs/symptoms of an infection. Clinic visits and/or sleep evaluations will be rescheduled to allow subject to be symptom-free of any type of systemic infection for at least 5 days.
4. Subject has uncontrolled hypertension (systolic blood pressure >160 mm Hg or diastolic blood pressure >100 mm Hg) at screening.
5. Subject has a known allergy or sensitivity to any ingredients in the study products.
6. Subject is a heavy consumer of caffeinated beverages (>400 mg caffeine/d from caffeine-containing products) within 2 weeks of screening.
7. Subject diagnosed with a psychiatric disorder that would impair their ability to perform the study, such as a psychotic disorder, bipolar disorder, neurodevelopmental disorder, post-traumatic stress disorder, etc. The subject should not currently be experiencing a major depressive episode. Psychiatric history will be assessed at screening then reassessed at the screening visit; In addition, the Mini International Neuropsychiatric Inventory will be conducted at the screening visit.
8. Subject has a history of use of psychotropic medications (including antidepressants, beta-blockers, and tranquilizers), stimulant medications, medical marijuana and/or narcotics within 4 weeks of screening.
9. Subject has used sleep aid medications, supplements, and/or products (over-the-counter or prescription), including antihistamines, within 2 weeks of screening. If use has occurred a wash-out period can be conducted.
10. Subject has a history of unconventional sleep patterns (e.g., night shift), chronic insomnia (defined as insomnia at least 3 d/week over the past month), a diagnosed sleep disorder (e.g., OSA), or a chronic medical condition that may impact energy/fatigue levels, in the judgment of the Investigator.
11. Subject has a history of cancer within 5 years prior to screening except for non-melanoma skin cancer.
12. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to use of a medically approved form of contraception throughout the study period.
13. Subject has a current or recent history (past 12 months of screening) or strong potential for drug or alcohol abuse. Alcohol abuse will be defined as > 14 drinks per week (1 drink = 12 oz. beer, 5 oz. wine, or 1.5 oz. hard liquor).
14. Subject has been exposed to any non-registered drug product within 30 d prior to screening.
15. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, might confound the interpretation of the study results, or put the person at undue risk.

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grandner, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Dept of Psychiatry Research facilities, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tubbs AS, Kennedy KER, Alfonso-Miller P, Wills CCA, Grandner MA. A Randomized, Double-Blind, Placebo-Controlled Trial of a Polyphenol Botanical Blend on Sleep and Daytime Functioning. Int J Environ Res Public Health. 2021 Mar 16;18(6):3044. doi: 10.3390/ijerph18063044. PMID 33809544

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred by self-referral, social media, and flyer advertising in Tucson, Arizona, USA.
Groups:
- Proprietary Spearmint Extract Blend: Subjects randomized into the active treatment group will be asked to consume 500 mg/day of the Proprietary Spearmint Extract Blend blend by mouth every night 30 mins before bed, complete a sleep diary upon waking and wear a Fitbit Charge 2 device for sleep monitoring for 30 days.
  A subset of this group will undergo 2 overnight polysomnography studies
  Proprietary Spearmint Extract Blend: Water extracted spearmint extract and green tea blend
- Control: Subjects randomized into the active treatment group will be asked to consume 500 mg/day of the excipient, microcrystalline cellulose by mouth every night 30 mins before bed, complete a sleep diary upon waking and wear a Fitbit Charge 2 device for sleep monitoring for 30 days.
  A subset of this group will undergo 2 overnight polysomnography studies
  Control: Placebo
Period: Overall Study
Arm/Group | Proprietary Spearmint Extract Blend | Control
Started | 53 | 52
Completed | 47 | 49
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — No longer eligible | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Final analyses included only 43 participants (4 excluded) in the active group, and 46 participants (3 excluded), due to missing data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Proprietary Spearmint Extract Blend | Control | Total
Number analyzed (Participants) | 43 | 46 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 46 | 89
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.91 (7.17) | 32.85 (8.62) | 31.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 54
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 33 | 36 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Asian | 0 | 8 | 8
  Race: Black or African American | 2 | 3 | 5
  Race: White | 30 | 25 | 55
  Race: Hispanic/Latino | 10 | 10 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 46 | 89

OUTCOME MEASURES:

1. Primary Outcome: Sleep Diary- Sleep Latency
Description: Time it takes to fall asleep after the lights have been turned off in minutes (Weekly averages)
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
minutes | -2.1 [-5.03 to .82] | -2.53 [-6.3 to 1.24]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — Significance set to 0.05; p = 0.1543, Paired T-test — The threshold for statistical significance was P< 0.05; Mean Difference (Net) = -2.1, 95% CI 2-sided [-5.03 to 0.82]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.1827, Paired T-test; Mean Difference (Net) = -2.53, 95% CI 2-sided [-6.3 to 1.24]

2. Primary Outcome: Fitbit - Rapid Eye Movement (REM) Sleep
Description: Change in Rapid Eye Movement (REM) Sleep in minutes (Weekly averages)
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
minutes | -0.2 [-1.96 to 1.56] | 1.58 [-0.77 to 3.94]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.8165, Paired T-test; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.96 to 1.56]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.1821, Paired T-test; Mean Difference (Net) = 1.58, 95% CI 2-sided [-0.77 to 3.94]

3. Secondary Outcome: Sleep Diary -Total Sleep Time
Description: Total Sleep Time in minutes
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
minutes | 20.94 [4.19 to 37.69] | 20.08 [-0.64 to 40.8]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.0156, Paired T-test; Mean Difference (Net) = 20.94, 95% CI 2-sided [4.19 to 37.69]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.0572, Paired T-test; Mean Difference (Net) = 20.08, 95% CI 2-sided [-0.64 to 40.8]

4. Secondary Outcome: Sleep Diary-Wake After Sleep Onset
Description: Number of awakenings after sleep onset
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: awakenings
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
awakenings | -4.48 [-9.37 to 0.41] | -3 [-8.1 to 2.1]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.0781, Paired T-test; Mean Difference (Net) = -4.48, 95% CI 2-sided [-9.37 to 0.41]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.242, Paired T-test; Mean Difference (Net) = -3.0, 95% CI 2-sided [-8.1 to 2.1]

5. Secondary Outcome: Sleep Diary- Sleep Efficiency
Description: ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed (percentage)
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
percent | 2.91 [0.49 to 5.32] | 4.66 [1.19 to 8.12]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.0195, Paired T-test; Mean Difference (Net) = 2.91, 95% CI 2-sided [0.49 to 5.32]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.0097, Paired T-test; Mean Difference (Net) = 4.66, 95% CI 2-sided [1.19 to 8.12]

6. Secondary Outcome: Sleep Diary - Objective Sleep Quality
Description: Sleep Quality (units on a visual analogue scale from 0-10, 0 being the worst outcome, 10 being the best outcome)
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
units on a scale | 0.93 [0.59 to 1.28] | 0.45 [0.08 to 0.81]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p < 0.0001, Paired T-test; Mean Difference (Net) = 0.93, 95% CI 2-sided [0.59 to 1.28]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.0179, Paired T-test; Mean Difference (Net) = 0.45, 95% CI 2-sided [0.08 to 0.81]

7. Secondary Outcome: Fitbit- Light Sleep
Description: Change in Light Sleep in minutes (Weekly averages)
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
minutes | -0.03 [-3.89 to 3.83] | -0.2 [-6.23 to 5.82]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.9875, Paired T-test; Mean Difference (Net) = -0.03, 95% CI 2-sided [-3.89 to 3.83]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.9463, Paired T-test; Mean Difference (Net) = -0.2, 95% CI 2-sided [-6.23 to 5.82]

8. Secondary Outcome: Fitbit - Total Sleep Time
Description: Total sleep time in minutes
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
minutes | 28.5 [9.84 to 47.17] | 9.84 [-15.63 to 35.31]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.0037, Paired T-test; Mean Difference (Net) = 28.5, 95% CI 2-sided [9.84 to 47.17]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — p<0.05; p = 0.4395, Paired T-test; Mean Difference (Net) = 9.84, 95% CI 2-sided [-15.63 to 35.31]

9. Secondary Outcome: Fitbit- Sleep Efficiency
Description: as for outcome 5
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
percent | -0.03 [-0.59 to 0.53] | -0.11 [-1.04 to 0.83]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.912, Paired T-test; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.59 to 0.53]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = .8207, Paired T-test; Mean Difference (Net) = -0.11, 95% CI 2-sided [-1.04 to 0.83]

10. Secondary Outcome: Fitbit- Deep Sleep
Description: Change in Deep Sleep in minutes (Weekly averages)
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
minutes | -0.89 [-2.26 to 0.47] | -0.24 [-3.35 to 2.86]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.1929, Paired T-test; Mean Difference (Net) = -0.89, 95% CI 2-sided [-2.26 to 0.47]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.8744, Paired T-test; Mean Difference (Net) = -.24, 95% CI 2-sided [-3.35 to 2.86]

11. Secondary Outcome: The Insomnia Severity Index (ISI)
Description: The Insomnia Severity Index (ISI): Total Score. Self-report rating scale assessing the severity of insomnia symptoms. Range 0-28 with higher scores indicating a more severe insomnia.
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
score on a scale | -0.95 [-2.45 to 0.54] | 0.96 [-0.5 to 2.42]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.2048, Paired T-test; Mean Difference (Net) = -.95, 95% CI 2-sided [-2.45 to 0.54]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.1933, Paired T-test; Mean Difference (Net) = 0.96, 95% CI 2-sided [-0.5 to 2.42]

12. Secondary Outcome: Sustained Attention
Description: Attentional lapses (failure to respond to stimuli within 500 ms) using the psychomotor vigilance test (PVT)
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: number of lapses
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
number of lapses | -1.69 [-3.25 to -0.13] | 0.41 [-0.88 to 1.71]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; change in mean number of lapses; Test type: Equivalence — P<0.05; p = 0.034, Paired T-test; Mean Difference (Net) = -1.69, 95% CI 2-sided [-3.25 to -0.13]
Statistical Analysis 2: Comparison: Control; Change in number of lapses; Test type: Equivalence — P<0.05; p = 0.5242, Paired T-test; Mean Difference (Net) = 0.41, 95% CI 2-sided [-0.88 to 1.71]

13. Secondary Outcome: Profile of Mood States (POMS)
Description: Profile of Mood States (POMS): Mood scores. The Profile of Mood States (POMS) is a psychological rating scale used to assess transient, distinct mood states. 65 adjectives rated on 5-point scale 0= not at all; 1=a little; 2=moderately; 3=quite a bit; 4=extremely. Factor analysis: 6 subscales tension-anxiety (9 items, score range: 0-36) depression (15 items, range 0-60) anger-hostility (12 items, range 0-48) vigor-activity (8 items, range 0-32) fatigue (7 items, range 0-28) confusion-bewilderment (7 items, range 0-28) Total mood disturbance (TMD) (range 0-200): TMD = (Tension + Depression + Anger + Fatigue + Confusion) - Vigour
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
score on a scale
  Total Mood Disturbance | 0.67 [-4.92 to 6.25] | 3.87 [-1.35 to 9.09]
  tension-anxiety | 0.05 [-1.11 to 1.21] | 1.54 [0.4 to 2.69]
  depression | 0.29 [-1.55 to 2.12] | 0.74 [-0.44 to 1.92]
  anger-hostility | 1.19 [-0.05 to 2.43] | 0.24 [-0.34 to 0.82]
  vigor-activity | 1.17 [-0.92 to 3.25] | -0.54 [-2.61 to 1.53]
  fatigue | 0.05 [-1.64 to 1.73] | 0.48 [-0.83 to 1.79]
  confusion-bewilderment | 0.26 [-0.65 to 1.18] | 0.33 [-0.5 to 1.15]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; POMS-TMD; Test type: Equivalence — P<0.05; p = 0.8106, Paired T-test; Mean Difference (Net) = 0.67, 95% CI 2-sided [-4.92 to 6.25]
Statistical Analysis 2: Comparison: Control; POMS-TMD; Test type: Equivalence — P<0.05; p = 0.1427, Paired T-test; Mean Difference (Net) = 3.87, 95% CI 2-sided [-1.35 to 9.09]
Statistical Analysis 3: Comparison: Proprietary Spearmint Extract Blend; POMS-Tension; Test type: Equivalence — P<0.05; p = 0.9344, Paired T-test; Mean Difference (Net) = 0.05, 95% CI 2-sided [-1.11 to 1.21]
Statistical Analysis 4: Comparison: Control; POMS-Tension; Test type: Equivalence — P<0.05; p = 0.0092, Paired T-test; Mean Difference (Net) = 1.54, 95% CI 2-sided [0.40 to 2.69]
Statistical Analysis 5: Comparison: Proprietary Spearmint Extract Blend; POMS-Depression; Test type: Equivalence — P<0.05; p = 0.755, Paired T-test; Mean Difference (Net) = 0.29, 95% CI 2-sided [-1.55 to 2.12]
Statistical Analysis 6: Comparison: Control; POMS-Depression; Test type: Equivalence — P<0.05; p = 0.2131, Paired T-test; Mean Difference (Net) = 0.74, 95% CI 2-sided [-0.44 to 1.92]
Statistical Analysis 7: Comparison: Proprietary Spearmint Extract Blend; POMS-Anger; Test type: Equivalence — P<0.05; p = 0.06, Paired T-test; Mean Difference (Net) = 1.19, 95% CI 2-sided [-0.05 to 2.43]
Statistical Analysis 8: Comparison: Control; POMS-Anger; Test type: Equivalence — P<0.05; p = 0.4117, Paired T-test; Mean Difference (Net) = 0.24, 95% CI 2-sided [-0.34 to 0.82]
Statistical Analysis 9: Comparison: Proprietary Spearmint Extract Blend; POMS-Fatigue; Test type: Equivalence — P<0.05; p = 0.9548, Paired T-test; Mean Difference (Net) = 0.05, 95% CI 2-sided [-1.64 to 1.73]
Statistical Analysis 10: Comparison: Control; POMS-Fatigue; Test type: Equivalence — P<0.05; p = 0.4649, Paired T-test; Mean Difference (Net) = 0.48, 95% CI 2-sided [-0.83 to 1.79]
Statistical Analysis 11: Comparison: Proprietary Spearmint Extract Blend; POMS-Confusion; Test type: Equivalence — P<0.05; p = 0.5656, Paired T-test; Mean Difference (Net) = 0.26, 95% CI 2-sided [-0.65 to 1.18]
Statistical Analysis 12: Comparison: Control; POMS-Confusion; Test type: Equivalence — P<0.05; p = 0.4307, Paired T-test; Mean Difference (Net) = 0.33, 95% CI 2-sided [-0.5 to 1.15]
Statistical Analysis 13: Comparison: Proprietary Spearmint Extract Blend; POMS-Vigor; Test type: Equivalence — P<0.05; p = 0.2651, Paired T-test; Mean Difference (Net) = 1.17, 95% CI 2-sided [-0.92 to 3.25]
Statistical Analysis 14: Comparison: Control; POMS-Vigor; Test type: Equivalence — P<0.05; p = 0.5992, Paired T-test; Mean Difference (Net) = -0.54, 95% CI 2-sided [-2.61 to 1.53]

14. Secondary Outcome: Perceived Stress Scale (PSS)
Description: Perceived Stress Scale (PSS): Total Score. The PSS is comprised of 14 items intended to measure how unpredictable, uncontrollable, and overloaded individuals find their life circumstances.Participants rate items on a 5-point Likert scale, ranging from 0 - "Never" to 4 - "Very often." Scores range from 0-56 higher scores indicate greater perceived stress.
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
score on a scale | 0.37 [-1.48 to 2.22] | 1.39 [-0.65 to 3.43]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.6869, Paired T-test; Mean Difference (Net) = 0.37, 95% CI 2-sided [-1.48 to 2.22]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.1769, Paired T-test; Mean Difference (Net) = 1.39, 95% CI 2-sided [-0.65 to 3.43]

15. Secondary Outcome: The Center for Epidemiological Studies Depression Scale (CESD)
Description: The Center for Epidemiological Studies Depression scale (CESD) Total score. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
score on a scale | 0.51 [-1.69 to 2.72] | 0.63 [-0.9 to 2.16]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.6422, Paired T-test; Mean Difference (Net) = 0.51, 95% CI 2-sided [-1.69 to 2.72]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.4106, Paired T-test; Mean Difference (Net) = 0.63, 95% CI 2-sided [-0.9 to 2.16]

16. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Pittsburgh Sleep Quality Index (PSQI): Total Score. The PSQI is a validated self-rating instrument assessing aspects of sleep quality.Minimum score 0 (better); maximum score 21 (worse) < or = 5 associated with good sleep quality; > 5 associated with poor sleep quality.
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
score on a scale | -0.23 [-1.05 to 0.58] | 0.11 [-0.77 to 0.99]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Test type: Equivalence — P<0.05; p = 0.5672, Paired T-test; Mean Difference (Net) = -0.23, 95% CI 2-sided [-1.05 to 0.58]
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — P<0.05; p = 0.805, Paired T-test; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.77 to 0.99]

17. Secondary Outcome: Sustained Attention
Description: Mean reaction time to stimuli using the psychomotor vigilance test (PVT)
Time Frame: Change from baseline after 30 days supplementation
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Proprietary Spearmint Extract Blend | Control
Number analyzed (Participants) | 43 | 46
milliseconds | -43.09 [-98.43 to 12.26] | -2.01 [-20.13 to 16.11]
Statistical Analysis 1: Comparison: Proprietary Spearmint Extract Blend; Change in lapse time; Test type: Equivalence — P<0.05; p = .1236, Paired T-test; Median Difference (Net) = -43.09, 95% CI 2-sided [-98.43 to 12.26]
Statistical Analysis 2: Comparison: Control; Change in lapse time; Test type: Equivalence — P<0.05; p = .8241, Paired T-test; Mean Difference (Net) = -2.01, 95% CI 2-sided [-20.13 to 16.11]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for approximately 1 month for each participant, as the duration of participation for any given participant was approximately 1 month.
Description: Any events of discomfort, pain, or abnormalities occurring during the course of the study.
Arm/Group | Proprietary Spearmint Extract Blend | Control
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 6/53 | 9/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proprietary Spearmint Extract Blend (N=53) | Control (N=52)
Stomach Discomfort (Gastrointestinal disorders) | 0 | 3 — Stomach discomfort symptoms.
Muscle pain (Musculoskeletal and connective tissue disorders) | 2 | 3 — Muscle pain or injury
Headache/migraine (General disorders) | 2 | 1 — Migraine/Headache
Sore throat (General disorders) | 2 | 1 — Sore or itchy throat
Tooth pain (General disorders) | 0 | 1 — Tooth pain or sensitivity
Ear ache (General disorders) | 1 | 0 — Ear ache
Sinus congestion (General disorders) | 1 | 1 — Sinus congestion
Fever (General disorders) | 1 | 0 — low-grade fever.
Fatigue (General disorders) | 1 | 0 — Weakness/fatigue

LIMITATIONS AND CAVEATS:
Models were not adjusted for baseline differences in race/ethnicity and REM sleep. Also, there is a lack of polysomnography data, which is the gold standard for evaluating sleep architecture, severely limits inferences on the effects of PBB on REM sleep. A further limitation is that neurocognitive testing was not conducted at a consistent time of day across individuals, meaning the results of neurocognitive testing could have been influenced by time-of-day testing effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT03567343/Prot_000.pdf